CLINICAL TRIAL: NCT04212468
Title: Home Blood Pressure Registration Study on Community Elderly Population(HOME Study)
Brief Title: Home Blood Pressure Monitoring Registration Study in the Elderly(HOME Study)
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018300H(R1)
Record Dates: First submitted 2019-12-24; First posted 2019-12-27 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Blood Pressure
Keywords: Blood Pressure; Elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples Without DNA — This study will collect 20 mL whole blood samples from subjects at one or more study visits. The whole blood will be processed to plasma and stored for testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
China is entering an aging society. As the number of elderly population continues to increase, the elderly are facing many social problems that deserve the attention of all sectors of society. Hypertension is one of the common diseases in the elderly population. Hypertension is the most common chronic diseases and a most important risk factor for cardiovascular and cerebrovascular diseases, and also a substantial public health problem. Home blood pressure monitoring is simple, not only can find hypertension, but also can guide the treatment of patients with hypertension. The purpose of the study is to investigate the association between home blood pressure and adverse outcomes in community elderly population.

DETAILED DESCRIPTION:
Study population includes subjects who living in community, of any race or ethnicity, 65 or older years of age, and have provided written informed consent to provide home blood pressure monitoring at one or more study visits.

Physical examination, questionnaire survey and biological sample collection will be conducted at baseline and the incidence of a composite of major adverse cardiovascular events will be investigated during follow-up.

ELIGIBILITY:
Inclusion Criteria:

•≥65 years old

* Signed informed consent
* Life expectancy is greater than 1 year

Exclusion Criteria:

* <65 years old
* Unsigned informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Study population includes subjects who living in community, of any race or ethnicity, 65 or older years of age.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | From date of inclusion until the date of death from any cause, assessed up to 1 year
  All-cause mortality was confirmed through a combination of hospital medical records, telephone contacts with patients or family members, and death registration at the Center for Disease Control and Prevention.
Cardiovascular Mortality | From date of inclusion until the date of death from any cause, assessed up to 1 year
  Cardiovascular mortality was defined as death attributable to an ischemic cardiovascular cause (including fatal cardiovascular events and stroke).

SECONDARY OUTCOMES:
Secondary outcomes of cardiovascular diseases | Through study completion, an average of 1 years
  The number of and the incidence rate of cardiovascular diseases.
Secondary outcomes of cerebrovascular diseases | Through study completion, an average of 1 years
  The incidence rate of cerebrovascular diseases.
Secondary outcomes of kidney | Through study completion, an average of 1 years
  The incidence rate of renal injure and end-stage renal disease
Secondary outcomes of hypertension | Through study completion, an average of 1 years
  The incidence rate of hypertension
Secondary outcomes of diabetes | Through study completion, an average of 1 years
  The incidence rate of diabetes

OTHER OUTCOMES:
Number of participants with reported hospitalization due to other diseases | From date of inclusion until the date of first event, assessed up to 1 year
  The incidence rate of tumor, fracture, cataract etc.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ying-qing, PhD, Study Chair — Guangdong Provincial People's Hospital
Locations (2):
- China (2):
  - Feng Yingqing, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No